CLINICAL TRIAL: NCT05497713
Title: Mindset Interventions to Facilitate Taking Cold Showers: A Randomized Controlled Study
Brief Title: Mindset Interventions to Facilitate Taking Cold Showers
Acronym: MICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jens Gaab (Other)
Responsible Party: Sponsor-Investigator, Jens Gaab, Sponsor-Investigator, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: eknz2022-00952
Record Dates: First submitted 2022-08-03; First posted 2022-08-11 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-03

CONDITIONS: Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Control Condition (No Intervention): No Mindset.
- Egoistic x Proximal (Experimental): Mindset: "This is my 5-minute exercise."
  Interventions: Other: Mindsets
- Egoistic x Distal (Experimental): Mindset: "I am doing this for my health."
  Interventions: Other: Mindsets
- Altruistic x Proximal (Experimental): Mindset: "I am saving one kilo of CO2: "
  Interventions: Other: Mindsets
- Altruistic x Distal (Experimental): Mindset: "I am doing this to fight climate change."
  Interventions: Other: Mindsets

INTERVENTIONS:
Other: Mindsets — The primary objective of this trial is to determine whether mindsets sustain the feasibility of taking cold showers over a 3-month period.
  Arms: Altruistic x Distal; Altruistic x Proximal; Egoistic x Distal; Egoistic x Proximal

SUMMARY:
The primary objective of this trial is to determine whether mindsets sustain the feasibility of taking cold showers over a 3-month period. Secondary objectives are to determine potential effects on physical and mental well-being, sleep quality, skin and hair appearance, perceived illness, and related sickness absences from work.

ELIGIBILITY:
Inclusion Criteria:

The investigators will include

* healthy participants between 18 and 65 years of age,
* which do not take cold shower on a regular basis.
* As there are no known gender differences, participants of both female and male sex are included.

Exclusion Criteria:

The investigators will exclude

* pregnant or lactating women by self-report and
* subjects with cardiac, pulmonary or any other severe disease by self-report.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-02-17 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Showering behaviour concerning frequency (Baseline) | Baseline
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning duration (Baseline) | Baseline
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning motivation (Baseline) | Baseline
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning frequency (Week 1) | Week 1
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning frequency (Week 2) | Week 2
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning frequency (Week 3) | Week 3
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning frequency (Week 4) | Week 4
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning frequency (Week 5) | Week 5
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning frequency (Week 6) | Week 6
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning frequency (Week 7) | Week 7
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning frequency (Week 8) | Week 8
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning frequency (Week 9) | Week 9
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning frequency (Week 10) | Week 10
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning frequency (Week 11) | Week 11
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning frequency (Week 12) | Week 12
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning duration (Week 1) | Week 1
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning duration (Week 2) | Week 2
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning duration (Week 3) | Week 3
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning duration (Week 4) | Week 4
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning duration (Week 5) | Week 5
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning duration (Week 6) | Week 6
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning duration (Week 7) | Week 7
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning duration (Week 8) | Week 8
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning duration (Week 9) | Week 9
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning duration (Week 10) | Week 10
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning duration (Week 11) | Week 11
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning duration (Week 12) | Week 12
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning motivation (Week 1) | Week 1
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning motivation (Week 2) | Week 2
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning motivation (Week 3) | Week 3
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning motivation (Week 4) | Week 4
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning motivation (Week 5) | Week 5
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning motivation (Week 6) | Week 6
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning motivation (Week 7) | Week 7
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning motivation (Week 8) | Week 8
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning motivation (Week 9) | Week 9
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning motivation (Week 10) | Week 10
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning motivation (Week 11) | Week 11
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning motivation (Week 12) | Week 12
  Participants will be asked their motivation for taking cold showers during the last week.

SECONDARY OUTCOMES:
WHO Five Well-Being Index | All secondary outcomes will be assessed at baseline and then monthly for 3 months.
  The WHO-5 is a short questionnaire designed to measure well-being. The WHO-5 consists of five questions. The answers are given on a six-level scale (0 - 5, where 0 represents "No time at all" and 5 "All the time"). The raw value is obtained by adding the answers. The raw value ranges from 0 to 25, where 0 is the lowest quality of life and 25 is the highest quality of life. The percentage value of 0 -100 is obtained by multiplying by 4. The percentage value 0 denotes the worst state of health, 100 the best. The processing time is less than one minute. Example: In the last 4 weeks I was happy and in a good mood.
Questionnaire for positive aspects of well-being in adults | All secondary outcomes will be assessed at baseline and then monthly for 3 months.
  The FEW 16 is a psychological self-evaluation procedure for the assessment of positive aspects of well-being in adults. The FEW 16 consists of 16 questions, of which 4 questions each are assigned to one of the following four scales: Ability to work under pressure, vitality, enjoyment, inner peace. The answers are given on a 6-level scale (1 - 6, where 6 represents "Does not apply at all" and 1 "Is absolutely true"). The processing time is estimated at five to ten minutes by adding up the 16 items you get an overall result between 16 - 96, whereas a lower overall result shows a higher physical wellbeing. Example: There's hardly anything that can upset me.
International Physical Activity Questionnaire | All secondary outcomes will be assessed at baseline and then monthly for 3 months.
  The IPAQ is a short questionnaire designed to measure physical activity. The IPAQ consists of six questions, of which 3 questions each are assigned to one of the following two scales: Strong physical exertion and light physical exertion. Either you have to tick an answer or you will be asked for a time in hours and minutes per week. The processing time is estimated at three minutes. Example: If you are thinking about physical activities where you are at least a little out of breath, such as running, hiking, dancing, gardening or many sports, how many days a week do you do physical activities of this kind?
Pittsburgh Sleep Quality Index | All secondary outcomes will be assessed at baseline and then monthly for 3 months.
  The PSQI is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete. The questionnaire offers seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totalling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. Example: How tired are you during the day?
Skin quality questionnaire | All secondary outcomes will be assessed at baseline and then monthly for 3 months.
  The SQQ is a short self-report questionnaire that assesses hand and skin quality. The measure consists of 4 items, whereas they measure appearance, intactness, moisture content and sensation on a 7-level scale (1-7), where higher scores denote a healthier quality of skin. The processing time is less than one minute each. Example: Appearance: Abnormal: redness, stains, rash. Normal: no redness, stains or rashes.
Sickness absence and illness days | All secondary outcomes will be assessed at baseline and then monthly for 3 months.
  Will be assessed at baseline and then monthly for 3 months. Participants are asked to retrospectively indicate the total number of days of absence from their work due to sickness and to indicate the number of days that they have had symptoms of illness, cold or flu during the last month. If participants indicate sickness absence or illness over five days, they are asked for the reason.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Gaab, Prof. Dr., Principal Investigator — University of Basel, Division Clinical Psychology and Psychotherapy
Locations (1):
- University of Basel Faculty of Psychology Division for Clinical Psychology and Psychotherapy, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No